CLINICAL TRIAL: NCT05328609
Title: An Exploratory Investigation of Dietary Supplementation and the Effect on Common Symptoms of Hormonal Imbalance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semaine Health (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20228Semaine
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Hormone Disturbance
MeSH Terms: conditions — Endocrine System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Semaine - The Daily
  Interventions: Dietary Supplement: Semaine Hormonal Imbalance & The Daily
- Control arm (No Intervention): No intervention for the time period

INTERVENTIONS:
Dietary Supplement: Semaine Hormonal Imbalance & The Daily — All participants will undergo a menstrual cycle without intervention to establish a baseline, and then will be given the intervention (dietary supplement) for a second menstrual cycle.
  Arms: Intervention arm

SUMMARY:
This is an open-label observational trial to study the effectiveness of a commercial dietary supplement and its effect on common symptoms of normal menstrual discomfort.

DETAILED DESCRIPTION:
This is an open-label observational trial to study the effectiveness of a commercial dietary supplement and its effect on common symptoms of normal menstrual discomfort.

It is hypothesized that the dietary supplement marketed as The Daily will improve subjective wellbeing in trial participants. It is further hypothesized that the dietary supplement will improve plasma biomarkers that have been previously correlated with insulin resistance.

A total of 45 participants will be recruited for the trial following screening, with the expectation that at least 35 will complete the trial. The trial will be fully remote, and all participants will undergo a menstrual cycle without intervention to establish a baseline, and then will be given the intervention (dietary supplement) for a second menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Female, aged 18-55 (roughly 75% 18-38 and 25% 45-55)
* Ability to take oral medication and be willing to adhere to the dietary supplement regimen (2 capsules per day)
* Willing to fast overnight (12+ hours) prior to the blood collection, and to perform an at-home fingerprick blood test
* Moderate self-reported discomfort related to perceived hormone imbalance. Participants must answer B or C on at least 3 of the following questions:

Exclusion Criteria:

* Current use of medication for high blood pressure or for blood thinning
* Diabetic, or on medication such as Metformin or Acarbose
* Pregnancy, breastfeeding, or attempting to become pregnant during study
* Known allergic reactions to components of the dietary supplement (sunflower oil, passionflower, berberine, or grape seed extract )
* Has exercised 3+ times per week of 30 minutes or more per session on average over the past 6 month
* On a ketogenic or vegan diet for more than the past 30 days
* If hormonal birth control, cannot stop during the duration of the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 45 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Discomfort associated with hormone imbalance | 60 days
  Changes in discomfort associated with the most common symptoms linked with perceived hormone imbalance. This outcome measure utilizes a questionnaire using the Likert scale (1-5) with lower values representing an improvement.

SECONDARY OUTCOMES:
Changes in biomarkers linked to insulin sensitivity | 60 days
  Changes in Hemoglobin A1C between baseline and intervention period.
Changes in biomarkers linked to metabolic regulation | 60 days
  Changes in HOMA-IR values between baseline and intervention period.

OTHER OUTCOMES:
Changes in perceived skin quality | 60 days
  Changes in perceived skin quality using skin images of participants' faces to compare changes between baseline and intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States